CLINICAL TRIAL: NCT04195204
Title: A Randomized, Double-blind, Placebo-controlled Pilot Trial Evaluating the Effect of Tropisetron on Prevention of Postoperative Cognitive Dysfunction in Patients After Cardiac Surgery
Brief Title: A Pilot Trial Evaluating the Effect of Tropisetron on Postoperative Cognitive Dysfunction After Cardiac Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Anshi Wu, Head of Anesthesiology, Beijing Chao Yang Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 29847819
Record Dates: First submitted 2019-11-27; First posted 2019-12-11 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2022-01

CONDITIONS: Postoperative Cognitive Dysfunction; Postoperative Delirium
MeSH Terms: conditions — Postoperative Cognitive Complications; Emergence Delirium | interventions — Tropisetron

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tropisetron (Experimental): Patients allocated to this arm will receive intravenous Tropisetron (5mg) before anesthesia induction and once daily for 7 days after surgery.
  Interventions: Drug: Tropisetron
- Placebo (Placebo Comparator): Patients allocated to this arm will receive an identical volume of normal saline before anesthesia and once daily for 7 days after surgery.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Tropisetron — Investigators administrated intravenously Tropisetron 5mg before anesthesia and once daily for 7 days after surgery.
  Arms: Tropisetron
Drug: Placebos — Investigators administrated intravenously saline solution as a placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the feasibility of a randomized, double-blind, placebo-controlled pilot trial evaluating the effect of tropisetron on prevention of postoperative cognitive dysfunction in patients after cardiac surgery.

DETAILED DESCRIPTION:
Postoperative cognitive dysfunction is a common complication during postoperative period，especially in elderly patients. It is characterized by cognitive decline, inattention and abnormal mental status following surgery. The presence of postoperative cognitive dysfunction is independently associated with poor recovery, increased hospital length of stay and increased mortality.

Tropisetron is a 5-HT3A receptor antagonist and is widely used to treat postoperative nausea and vomiting. Previous studies found that tropisetron has positive effect on cognitive function.

We have designed a randomized, double-blind, placebo-controlled trial to determine if tropisetron has a positive effect on postoperative coginitive function in patients after cardiac surgery. Several assessements which are related to delirium, cognitive function, sleep and functional status, blood sample collection and EEG recordings will be involved in the trial. Moreover, we have assumed a few long-term follow-ups.

Given the complexity of the trial, we have decided to implement a pilot trial to assess the feasibility and provide vital data for future formal trial.

ELIGIBILITY:
Inclusion Criteria:

1. Written consent given
2. Scheduled to undergo elective coronary artery bypass graft surgery under general anesthesia
3. ASA Physical Score I-IV

Exclusion Criteria:

1. Inability to give informed consent.
2. Contraindications to tropisetron.
3. Critical preoperative state, including preoperative left ventricular ejection fraction less than 30%, ventricular tachycardia or ventricular fibrillation, preoperative cardiopulmonary resuscitation, preoperative intra-aortic balloon pump (IABP) or mechanical circulatory requirement.
4. History of neuropsychiatric diseases (such as dementia, epilepsy, Parkinson's disease, or schizophrenia).
5. History of antipsychotic drug use.
6. Pre-existing severe cognitive impairment at baseline, defined as a Montreal Cognitive Assessment (MoCA) score below 10

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
The feasibility of tropisetron intervention on POCD in patients after cardiac surgery | Within 30 days after surgery
  The feasibility will mainly be determined by the percentage of participants who completed the whole study procedure from recruitment to the 1-month follow-up.

SECONDARY OUTCOMES:
Incidence of postoperative cognitive dysfunction | One day before surgery, discharge from hospital and 1 month after surgery
  Screening of the patients regarding a POCD by Repeatable Battery Neuropsychological Status (RBANS). Besides, the changes in SCWT and IRI scores will be an additional indication of POCD.
Incidence of postoperative delirium | Within 7 days after surgery
  Screening of the patients regarding a postoperative delirium by The Confusion Assessment Method for The Intensive Care Unit (CAM-ICU)
Functional status measurement | One day before surgery and 1 month after surgery
  Screening of the patients by Barthel Index scale ranging from 0 to 100, where less than 20 indicates total dependence, 20-35 scores indicate severe dependence, 40-55 scores indicate moderate dependence, equal or over 60 indicates mild dependency and 100 indicates independence.
EEG frequency spectrum | Within 3 days after surgery
  Electroencephalography will be recorded at different points of time as follows and EEG characteristics including power in alpha, beta, theta, delta, gamma, spectrum will be extracted using MATLAB:
  1. before anesthesia introduction
  2. during anesthesia
  3. 1 day after surgery
  4. 2 days after surgery
  5. 3 days after surgery
Postoperative Pain | Within 7 days after surgery
  Visual Analogue Scale will be used to assess postoperative pain of patients. Numerical rating scale ranging from 0 to 10, where 0 indicates no pain and 10 indicates the worst pain.
Sleep Quality | Within 30 days after surgery
  Sleep diary and subjective sleep quality scores（Visual Analogue Scale） will be used to assess postoperative sleep quality of patients within 7 days after surgery.
  Chinese version of the Pittsburgh sleep quality index (PSQI) will be used to assess sleep quality and disturbances. Nineteen individual items generate seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for these seven components yields one global score. The total score is between 0 and 21. The total score ≤ 5 indicates good sleep quality，> 5 indicates poor sleep quality. PSQI will be recorded at different points of time as follows：
  1. 1 day before surgery
  2. 30 days after surgery
Incidence of postoperative nausea and vomiting | Within 7 days after surgery
Length of ICU stay | From the date of admission until discharged from ICU, up to 30 days
Length of Hospital stay | From the date of admission until discharged from hospital, up to 30 days
Incidence of major adverse cardiac and cerebral events | Within 30 days after surgery
  MACCE comprises all-cause mortality, myocardial infarction, repeat unplanned revascularization (surgical revision or percutaneous transluminal coronary angioplasty), and stroke
Inflammatory biomarkers | Within 7 days after surgery
  lood samples will be collected at different points of time as follows:
  1. before anesthesia introduction
  2. 1 day after surgery
  3. 3 days after surgery
  4. 7 days after surgery Levels of serum biomarkers, including but not limited to, interleukin (IL)-1β, IL-6, IL-8, tumor necrosis factor (TNF)α, Interferon (IFN)γ, Tau, vascular endothelial growth factor (VEGF)D and brain-derived neurotrophic factor (BDNF) will be examined using these specimens

OTHER OUTCOMES:
Incidence of major adverse cardiac and cerebral events | Within 30 days after surgery
  Other adverse events within 30 days after surgery were noted

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Chaoyang Hospital, Capital Medical University, Beijing, China